CLINICAL TRIAL: NCT04745039
Title: Guo's Entry Tear Repair :The First in Man Study of Endopatch System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endopatch V1.0
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-02

CONDITIONS: Chronic Stanford B Type Aortic Dissection Proximal Tear

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endopatch System (Experimental): Participants will be treated with Endopatch System
  Interventions: Device: Endopatch System

INTERVENTIONS:
Device: Endopatch System — The patch system for aortic dissection tear is composed of a dissection tear patch system and an adjustable bend conveyor. The patch system is composed of a patch and a conveying steel cable. The patch is pre-installed on the conveying steel cable.

SUMMARY:
A prospective, single-center, first in man study to evaluate the safety and efficacy of Endopatch System manufactured by Hangzhou Endonom Medtech Co., Ltd. for the Chronic Stanford B type aortic dissection proximal tear.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old, no gender limitation;
2. Able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the patient him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol;
3. Diagnosed as chronic Stanford type B aortic dissection;
4. Maximum diameter of the intimal tears is between 2mm and 20mm;
5. Important branch vessels will not be covered after intimal tears closure;
6. Aortic endovascular treatment can be performed with appropriate arterial access.

Exclusion Criteria:

1. Diagnosed as acute, subacute aortic dissection;
2. Intermural hematoma, aortic ulcer, pseudoaneurysm, and severe aortic calcification;
3. The minimum distance between the intimal tears of the aortic intimal flaps and the root of the intimal flaps is less than the radius of the patch to be used (the patch cannot be deployed flat);
4. Pregnant, breastfeeding or cannot contraception during the trial period;
5. Participated in clinical trials of other drugs or devices during the same period;
6. The same operation requires intervention in other vascular diseases (such as coronary artery, renal artery, superior mesenteric artery, etc.), and the postoperative drug treatment plan is therefore affected;
7. Allergic to contrast agents, anesthetics, patches, and delivery materials;
8. Cannot tolerate anesthesia;
9. Severe liver, kidney, lung, and heart function abnormalities before surgery [Serum creatinine exceeds 2 times the upper limit of normal; Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeds 5 times the upper limit of normal; Serum total bilirubin (STB) more than 2 times the upper limit of normal; Left ventricular ejection fraction is lower than normal by cardiac color Doppler ultrasound examination];
10. History of myocardial infarction, TIA or cerebral infarction within the past 3 months;
11. Life expectancy is less than 12 months (such as advanced malignant tumors)
12. Acute systemic infection
13. Investigator judged that not suitable for interventional treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
No major adverse events within 30 days after surgery. | 30 days after operation
  Major adverse events within 30 days after operation refer to all-cause death, myocardial infarction, ischemic stroke, respiratory failure, liver failure, renal failure, intestinal necrosis, paraplegia, and amputation within 30 days after operation. Among them, renal failure refers to long-lasting dialysis, kidney transplantation, or other fatal results. Intestinal necrosis is intestinal ischemia that requires bowel resection or other fatal consequences. Severe lower limb ischemia refers to new severe limp or resting pain after surgery.
The success rate of entry tears closure 6 months after operation. | 6 months after operation
  The success rate of intimal tears closure at 6 months is a composite index, including immediate technical success after the operation and no leakage of the intimal tears sealed by the DSA 6 months after the operation, no displacement of the patch, and no second occurrence during the follow-up period.

SECONDARY OUTCOMES:
All-cause mortality, aortic dissection-related mortality, serious adverse events, and device-related adverse events. | 30 days, 6 months, and 12 months after operation
  1. All-cause mortality 30 days, 6 months, and 12 months after operation;
  2. Mortality related to aortic dissection 30 days, 6 months, and 12 months after operation;
  3. Incidence of serious adverse events 30 days, 6 months, and 12 months after operation;
  4. Incidence of device-related adverse events 30 days, 6 months, and 12 months after operation.
False lumen thrombosis of the descending thoracic aorta 1 month, 6 months, 12 months after operation | 1 month, 6 months, 12 months after operation
  False lumen thrombosis of the descending thoracic aorta 1 month, 6 months, 12 months after operation.
Change of false lumen diameter in descending thoracic aorta 1 month, 6 months, 12 months after operation | 1 month, 6 months, 12 months after operation
  Change of false lumen diameter in descending thoracic aorta 1 month, 6 months, 12 months after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ge YY, Zhang HP, Guo W. A Novel Endovascular Double-Disc Implant for Sealing Intimal Tears in Aortic Dissection. JACC Asia. 2023 Nov 21;3(6):937-941. doi: 10.1016/j.jacasi.2023.09.009. eCollection 2023 Dec. PMID 38155784